CLINICAL TRIAL: NCT05907083
Title: Sexual Dimorphism of Sphenoid and Maxillary Air Sinuses Via 3D Volumetric Segmentation of CBCT: A Cross Sectional Study
Brief Title: Sexual Dimorphism of Sphenoid and Maxillary Air Sinuses Via 3D Volumetric Segmentation of CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ehab Samir Ali Abuelola, PhD Candidate, Cairo University
Other Study IDs: ORAD7 -1 -1
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Sexual Dimorphism; Cone-beam Computed Tomography; Maxillary Sinus; Sphenoid Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult CBCT Scan: CBCT Radiation
  Interventions: Radiation: cone beam computer tomography

INTERVENTIONS:
Radiation: cone beam computer tomography — Cone Beam CT Radiation
  Other Names: CBCT

SUMMARY:
Sexual dimorphism from skeletal remains a crucial step towards biological profile reconstruction since these are some of the last structures to remain after death. Paranasal sinuses remain intact even in extreme situations and are able to resist adverse environmental conditions due to their unique properties. The maxillary sinus is the largest of all paranasal sinuses and is considered as characteristic entity like human fingerprints for each person. Also, sphenoid air sinus is located deeply in the skull and is enveloped by different structures inside the sphenoid body. It is the least possibly affected by external deteriorating factors. Owing to limited research on the Egyptian population on the role of 3D volumetric assessment of paranasal sinuses in forensics, this study will be designed to investigate the significance of the volume of both sphenoid and maxillary sinuses in sexual discrimination.

DETAILED DESCRIPTION:
Sexual dimorphism from skeletal remains a crucial step towards biological profile reconstruction since these are some of the last structures to remain after death. Paranasal sinuses remain intact even in extreme situations and are able to resist adverse environmental conditions due to their unique properties. The maxillary sinus is the largest of all paranasal sinuses and is considered as characteristic entity like human fingerprints for each person. Also, sphenoid air sinus is located deeply in the skull and is enveloped by different structures inside the sphenoid body. It is the least possibly affected by external deteriorating factors. Owing to limited research on the Egyptian population on the role of 3D volumetric assessment of paranasal sinuses in forensics, this study will be designed to investigate the significance of the volume of both sphenoid and maxillary sinuses in sexual discrimination.

* CBCT Scans included in this study performed using CBCT machine (Planmeca Promax 3D MID (Planmeca OY, Helsinki, Finlan.
* Exposure parameters of the scans will vary depending on patients' sizes (according to the manufacturer's recommendations).
* Full maxillofacial scans with 0.4 voxel sizes will be reviewed.
* DICOM files of CBCT images will be analysed using Mimics software (version 21.0; Materialize, Leuven, Belgium).
* To measure volumes of the sphenoid and maxillary sinuses, Semiautomatic segmentation will be done using the new mask tool in Mimics software, thresholding will be applied to optimize sinus segmentation.
* The region-growing tool will be used on the previous mask to exclude any data not related to the sinuses and ensure the segmentation precision. Mask calculation will be done and the segmented sinus will be calculated as 3D Volume.
* The volume will be measured in cubic millimeters (mm3) by the software itself.
* The segmentation process will be carried out by one radiologist with 10 years of experience. For inter-observer agreement 50 cases will be segmented again by another radiologist with 15 years of experience in a separate session. Also, the analysis of data will be reviewed by both of them separately.
* CBCT images will be coded and radiologists will be blinded from the age and sex of patients and from the other observers' readings.
* Interpretation will be based mainly on software's segmentation capabilities minimizing the operator's skill dependence.

ELIGIBILITY:
Inclusion Criteria:

* Adult Egyptian patients
* Both sexes of age 20 to 60
* Normal complete upper dental arch
* Normal anatomy of the studied air sinuses.

Exclusion Criteria:

* Scans with any facial pathosis like (tumors, odontogenic lesions, and bone lesions).
* Scans showing any skeletal asymmetries, craniofacial traumas and developmental anomalies such as palatal cleft.
* Patients with fractures or lesions affecting the studied sinuses.
* Scans with insufficient Field of view
* Scans of low-resolution quality.
* Presence of considerable artifacts.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: CBCT maxillofacial scans belonging to Egyptian individuals will be examined
Sampling Method: Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Sexual dimorphism of maxillary air sinuses via volumetric segmentation | 1 year

SECONDARY OUTCOMES:
Sexual dimorphism of Sphenoid sinuses via volumetric segmentation | 1 year
Determination of age via sphenoid and maxillary air sinuses volumetric segmentation | 1 year